CLINICAL TRIAL: NCT05982158
Title: Remotely Delivered Avatar-mediated Therapy Versus Cognitive Behavioural Therapy for Persisting Auditory Hallucinations: Randomised Controlled Superiority Trial
Brief Title: Avatar-mediated Therapy Versus Cognitive Behavioural Therapy for Persisting Experiences of Hearing Voices
Acronym: AMETHYST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Swinburne University of Technology (Other)
Collaborators: University of Copenhagen (Other); University of Manchester (Other); University of Melbourne (Other); Monash University (Other); Perth Voices Clinic (Unknown); University of the Sunshine Coast (Unknown); University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GNT2015133
Record Dates: First submitted 2023-07-20; First posted 2023-08-08 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Auditory Hallucination; Psychotic Disorders; Schizophrenia and Related Disorders
Keywords: Auditory verbal hallucinations; Psychosis; Schizophrenia; Psychological therapy; Cognitive behavior therapy; Avatar therapy; Virtual reality; Telehealth
MeSH Terms: conditions — Hallucinations; Psychotic Disorders; Schizophrenia | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: AMETHYST is a pragmatic, parallel group, randomised controlled superiority trial, comparing avatar therapy to CBT for persisting AVHs, with the primary outcome of post-intervention hallucination severity. In both arms, therapy will be delivered within a three-month period, with assessor-blinded assessments completed at baseline, post-intervention (3 months), and follow-ups (6 months and 9 months).
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors involved in completing the assessments will be masked to treatment condition. Due to the type of intervention, it will not be possible to blind therapists delivering the interventions to participant's treatment condition. Clinicians providing routine care will also be aware of the condition. Participants will be instructed not to discuss treatment with their outcomes assessor. When an interview leads to unblinding, the outcomes assessor will be replaced.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioural Therapy (CBT) (Active Comparator): The standard therapy arm will be based on a focused cognitive behavioural therapy (CBT) protocol for AVHs. Sessions will involve discussing the characteristics of participant's AVHs, before applying core CBT approaches, adapted to the AVH experience, to conduct a thorough cognitive behavioural assessment with a focus on coping strategy enhancement and cognitive restructuring.
  Interventions: Behavioral: Cognitive behavioural therapy (CBT)
- Avatar Therapy (Experimental): The experimental arm will use avatar therapy. Sessions will involve generating an audio-visual avatar as a virtual representation of the primary 'voice' that the participant hears. This will be used to recreate AVHs experientially and allow participants to practice alternative ways of responding to the 'voice'. This innovative approach will be combined with the use of broader CBT methods.
  Interventions: Behavioral: Avatar therapy

INTERVENTIONS:
Behavioral: Avatar therapy — Seven 50-minute therapy sessions conducted by videoconferencing.
  Arms: Avatar Therapy
Behavioral: Cognitive behavioural therapy (CBT) — Seven 50-minute therapy sessions conducted by videoconferencing.
  Arms: Cognitive Behavioural Therapy (CBT)

SUMMARY:
The aim of this study is to compare the effects of a new psychological therapy, Avatar Therapy, to the current standard therapy, Cognitive Behavioural Therapy (CBT), in improving outcomes in people living with psychotic disorders who have persisting experiences of hearing voices (auditory verbal hallucinations, AVHs).

DETAILED DESCRIPTION:
Continually hearing critical, abusive or threatening voices (auditory verbal hallucinations, AVHs) is a major persisting and disabling symptom of psychotic disorders such as schizophrenia. Current treatments have universally had only modest impact. In preliminary trials, a brief digitally supported treatment, using avatars to recreate AVHs during therapy, has produced some of the largest reductions in AVH severity seen to date. To definitively test the superiority of this innovative treatment, AMETHYST is a randomised controlled trial comparing avatar therapy to current recommended best practice treatment, CBT, for medication-resistant AVHs.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia-related disorder or a mood disorder with psychotic symptoms diagnosis confirmed using the Structured Clinical Interview for DSM (SCID)
* Experiencing current auditory verbal hallucinations as measured by the Positive and Negative Syndrome Scale (PANSS) item P3 ≥ 4
* Auditory verbal hallucinations present for at least one year
* AVHs include significant negative content (PSYRATS item 6 ≥ 2) and/or AVHs are distressing (PSYRATS item item 9 ≥ 2)
* Current treatment with antipsychotic medication, or has been treated with antipsychotic medication in the past, with at least two different antipsychotic compounds, and these have been discontinued due to insufficient treatment response and/or poor tolerability.
* Access to the internet and a computer or other device on which videoconferencing software can be used
* Sufficient fluency in English for meaningful participation
* Age 18 or over
* Ability to give informed consent

Exclusion Criteria:

* Auditory verbal hallucinations attributable to a primary substance use disorder or organic disorder
* Estimated full scale IQ < 70 (using the Test of Premorbid Functioning, TOPF)
* Within the last month or planned at the time of intake: a change of antipsychotic medication,
* Current or within the past 3 months receipt of individual psychological therapy for hearing voices, or receipt of electro-convulsive therapy or other brain stimulation treatment;
* AVHs in a language not spoken by the therapists.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2023-08-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Auditory verbal hallucination severity, measured by total score on the Psychotic Symptom Rating Scale - Auditory Hallucinations Scale (PSYRATS-AHS) | Immediately post intervention (3 months), controlling for baseline
  Clinician-rated scale providing an index of overall severity based on 11 aspects of hallucinations (frequency, duration, intensity of distress, etc.), rated masked to treatment allocation. Each of the 11-items are scored on a 5-point scale (0 - 4), scores range from 0 to 44, with increased symptom expression indicated by higher scores.

SECONDARY OUTCOMES:
Change in auditory verbal hallucination severity, measured by total score on the Psychotic Symptom Rating Scale - Auditory Hallucinations Scale (PSYRATS-AHS) over follow-ups | Baseline, follow-ups (6 and 9 months)
  Follow-up timepoints on the clinician rated scale that is used to measure the primary outcome. Includes 11-items that are scored on a 5-point scale (0 - 4), scores range from 0 to 44, with increased symptom expression indicated by higher scores.
Change in auditory verbal hallucination-related distress, measured by the Psychotic Symptom Rating Scale - Auditory Hallucinations Scale (PSYRATS-AHS) Distress Score | Baseline, immediately post intervention (3 months), and follow-ups (6 and 9 months)
  Subscale of the clinician-rated scale that is used to measure the primary outcome. This includes 1-item that is scored on a 5-point scale (0 - 4), score ranges from 0 to 4, with increased symptom expression indicated by a higher score.
Remission of hallucinations, indexed by a score below 3 on the Hallucination scale of the Positive and Negative Syndrome Scales (PANSS) | Immediately post intervention (3 months), follow-ups (6 and 9 months)
  Clinician-rated scale to assess presence and severity of hallucinations. This includes 1-item, scored from 1 to 7, with increased symptom expression indicated by higher scores.
Change in overall psychosis symptom severity, measured by Positive and Negative Syndrome Scales (PANSS) total and sub scale scores | Baseline, immediately post intervention (3 months), follow-ups (6 and 9 months)
  Clinician-rated scale to assess overall psychotic symptom severity on total and sub scale scores (Positive, Negative and General Psychopathology). Includes a total of 30-items that are scored on a 7-point scale (1 - 7). Total score ranges from 30 to 210; Positive and Negative sub scale scores range from 7 to 49; General Psychopathology sub scale scores range from 16 to 112. Higher scores are indicative of increased symptom expression.
Change in depressive symptoms, measured by the Calgary Depression Scale for Schizophrenia (CDSS) | Baseline, immediately post intervention (3 months), follow-ups (6 and 9 months)
  Clinician-rated scale to assess depressive symptoms in schizophrenia. Includes a total of 9-items that are scored on a 4-point scale (0 - 3). Total score ranges from 0 to 27, with higher scores indicative of increased symptom expression.
Change in anxiety symptoms, measured by the anxiety scale of the 21-item Depression Anxiety Stress Scale (DASS-21) | Baseline, immediately post intervention (3 months), follow-ups (6 and 9 months)
  Self-report measure to assess depression, anxiety, and stress. Includes a total of 21-items that are scored on a 4-point scale (0 - 3). Scoring is made up of three sub scales that each include 7 items (Depression, Anxiety, and Stress). The scores for each of the three sub scales range from 0 to 42, with higher scores indicating increased symptom expression.
Personal recovery (consumer-defined recovery), measured by the Questionnaire for the Process of Recovery (QPR) | Baseline, immediately post intervention (3 months), follow-ups (6 and 9 months)
  A self-report measure to assess consumer-defined recovery from psychosis. Includes 15-items that are rated on a 5-point scale, scores range (0-4), scores range from 0-60, with greater recovery indicated by higher scores.

OTHER OUTCOMES:
Satisfaction with therapy, measured by the Client Satisfaction Questionnaire (CSQ-8) | Immediatedly post-intervention (3 months)
  The 8-item Client Satisfaction Questionnaire (CSQ-8) will be administered at the end of treatment to assess and compare participants satisfaction across the two therapies. In addition, a group of participants will be purposively sampled to be invited to take part in a detailed semi-structured qualitative interview (conducted by a non-blinded researcher) about their experiences of the intervention.
Adverse effects of therapy | Immediately post-intervention (3 months)
  Negative psychological effects such as discomfort and anxiety that are relevant to tolerability will be measured using the Negative Effects Questionnaire (NEQ), a 32-item psychometrically validated questionnaire developed for monitoring adverse effects of psychological therapies. The NEQ items are scored on a 5-point Likert scale (0-4) and differentiates between negative effects attributed to treatment and those caused by other circumstances. Potential deterioration in AVHs will be reported for each group by the proportion of participants showing deterioration above a reliable change index for the PSYRATS. Serious adverse events (SAEs) will include participant death, hospital admissions, episodes of crisis, assessment team treatment, attempted suicide, and violent incidents leading to police involvement; these will be recorded systematically.
Cost-effectiveness | Immediately post intervention (3 months), follow-ups (6 and 9 months)
  Cost-effectiveness calculations will use the Assessment of Quality of Life - 8 Dimensions (AQoL-8D) to measure quality of life as an index of utility, expressed in quality-adjusted life years (QALYs). The AQoL-8D includes 35-items covering 8 dimensions: Independent Living, Pain, Senses, Mental Health, Happiness, Coping, Relationships, and Self-worth. To both measure treatment as usual (TAU) and determine broader treatment costs, a Resource Use Questionnaire (RUQ), adapted for use in this population, will be used. Consent for administrative data (e.g., Medicare and Pharmaceutical Benefits, MBS/PBS) will also be collected. Prescribed medication will be considered in terms of both cost and chlorpromazine -equivalent antipsychotic medication dose.
Change in the impact of AVHs, measured by the Voice Impact Scale (VIS) | Baseline, immediately post-intervention (3 months), follow-ups (6 and 9 months)
  Self-report measure of the degree of impact of hearing voices on domains of distress, interference with day-to-day functioning, and positive impacts. Includes 24-items. Each item is individually scored from 0 (disagree completely) to 10 (agree completely) with higher scores on individual items indicating higher agreement with the items listed experience. Not applicable is also available if the item is not relevant.
Change in AVH content, measured by the Voice Content Questionnaire (VCQ) | Baseline, immediately post-intervention (3 months), follow-ups (6 and 9 months)
  Self-report process measure of the degree of negative and positive content of auditory verbal hallucinations. Includes 20-items scored on a 5-point rating scale (0 - 4). Two subscales are created: Positive and Negative sub scales with scores for each ranging from 0 to 40. Higher scores indicate increasing symptom expression of either positive or negative content.
Change in attention paid to AVHs, measured by the Listening and Believing Assessment for Voices | Baseline, immediately post-intervention (3 months), follow-ups (6 and 9 months)
  Self-report process measure of the extent to which the person listens to and believes AVH content. Each of the 18-items are scored on a 4-point scale (0-3), with items divided between four subscales: Actively listening to nasty voices, passively listening to nasty voices, believing nasty voices, and disregarding nasty voices. Scores for the first three respective subscales range from 0-12 and scores range from 0-20 for the disregarding nasty voices sub scale. Higher scores are indicative of greater engagement in sub scale listening and believing activities.
Change in confidence in coping with AVHs - single item rating | Baseline, immediately post-intervention (3 months), follow-ups (6 and 9 months)
  Self-report process measure. One-item scored on a scale from 1 - 10, with increasing confidence indicated by higher scores.
Change in interpersonal appraisals of AVHs, measured by the Beliefs About Voices Scale (BAVQ-R) | Baseline, immediately post-intervention (3 months), follow-ups (6 and 9 months)
  Self-report process measures of interpersonal appraisals of AVHs (e.g., as malevolent or powerful). Includes 18-items that are scored on a 4-point scale (0-3), with scores ranging from 0-18 for each of the three sub scales: malevolence (6-items), benevolence (6-items), and omnipotence (6-items). Greater malevolent, benevolent or omnipotent beliefs about voices are indicated by higher scores on each of their respective sub scales.
Change in interpersonal appraisals of AVHs, measured by the Voice Power Differential Scale (VPDS) | [Time Frame: Baseline, immediately post-intervention (3 months), follow-ups (6 and 9 months)]
  Self-report process measures of interpersonal appraisals of AVHs (e.g., as malevolent or powerful). Includes 7-items measuring the power differential between the voice and voice hearer on dimensions including, power, strength, confidence, respect, ability to inflict harm, superiority and knowledge that are each scored on a 5-point scale (1-5), with scores ranging from 7 to 35. Higher scores indicate greater perceived power differential in favour of the voice.
Change in interpersonal responses to AVHs, measured by the APPROVE | Baseline, immediately post-intervention (3 months), follow-ups (6 and 9 months)
  Self-report process measure of assertive, aggressive and passive interpersonal responses to AVHs. Includes 15-items that are scored on an 11-point scale (0-10), scores range from 0-150, with items divided between three sub scales: one assertive responding sub scale (5-items) and two non-assertive responding sub scales (passive and aggressive; 5-items each). Higher scores on each sub scale are indicative of greater engagement in sub scale behaviours.
Change in flexibility in interpersonal reponse to AVHs, measured by the Circumplex Scales for Interpersonal Efficacy (CSIE) | Baseline, immediately post-intervention (3 months), follow-ups (6 and 9 months)
  Self-report process measure of self-efficacy to respond in a range of different ways in a relationship, adapted to rate responses to AVH. Includes a total of 32-items that are scored from 0 (not at all confident) to 10 (absolutely confident). Eight sub scales (Agnetic, Agnetic & Uncommunal, Uncommunal, Unagnetic & Uncommunal, Unagnetic, Unagnetic & Communal, Communal, Agnetic & Communal) each of which include 4-items are calculated. The score of each sub scale is the sum of the 4-items (ranging from 0 to 40) divided by 4. Higher scores indicate increasing confidence.
Change in positive and negative views of self and others, measured by the Brief Core Schema Scales (BCSS) | Baseline, immediately post-intervention (3 months), follow-ups (6 and 9 months)
  Self-report process measure. Includes 24-items that are scored on a 5-point scale (0 - 4), scores range from 0 to 96, with four sub scales: negative-self, positive-self, negative others, and positive-others. Each sub scale includes 6-items, scores range from 0-24, with stronger belief in schemas indicated by higher scores.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Thomas, Principal Investigator — Swinburne University of Technology
Locations (1):
- Swinburne University of Technology, Hawthorn, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No